CLINICAL TRIAL: NCT02600416
Title: Effects of AV Port Reversal in Citrate CVVH - The CIRE Study (CItrate REcirculation Study)
Brief Title: The CIRE Study (CItrate REcirculation Study)
Acronym: CIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Willem Boer, MD, Ziekenhuis Oost-Limburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIRE study
Record Dates: First submitted 2015-10-15; First posted 2015-11-09 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AV port reversal (Other): Patients undergoing citrate CVVH.
  Interventions: Other: AV port reversal

INTERVENTIONS:
Other: AV port reversal — Reversal of the AV port at 1h Reversal of the AV port to start position at 7h

SUMMARY:
The aim of this study is to determine the effects of AV port reversal (AVPR) on recirculation, clearance, post-filter ionized calcium and subsequently citrate dosing.

DETAILED DESCRIPTION:
Rationale:

AV port reversal (AVPR) has been demonstrated to increase recirculation in venous catheters used in ICU for CVVH. The effects of this frequently used manoeuvre have not been described in the setting of CVVH using regional citrate anticoagulation.

Objective:

The aim of this study is to determine the effects of AVPR on recirculation, clearance, post-filter ionized calcium and subsequently citrate dosing.

Study design and methods:

Open trial studying the effect of AVPR in patients undergoing citrate CVVH. After measurement in standard catheter configuration, AVPR is performed after which effects on catheter recirculation, clearance, citrate dosing and post-filter ionized calcium (iCa) are monitored.

Sample sites:

Arterial line, arterial (pre-filter) port, postfilter port (after postdilution and calcium compensation), effluent sample. All flow rates to be noted.

Study population:

Twelve patients admitted to intensive care, requiring continuous renal replacement therapy (CRRT) for AKI. Patients are preferably anuric and have achieved good metabolic control under CVVH before inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients requiring CRRT for AKI (RIFLE criteria)
* Written informed consent from the patient or legal representative
* No AV port reversal had taken place before inclusion in the study
* Diuresis is minimal or the patient is anuric so that effects of changes in clearance as a consequence of diuresis are minimalized and do not influence study outcomes.
* The patient has undergone CVVH for a number of days, ensuring good metabolic control, so that possible short term loss of clearance as a consequence of AV port reversal has no detrimental effects.

Exclusion Criteria:

* pre-existing chronic renal insufficiency requiring dialysis
* chronic immunosuppression
* liver cirrhosis Child-Pugh C
* severe or shock-related hepatitis
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-12; Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
change in citrate concentration in circuit after AV port reversal | 8 hours
change in post-filter ionised Ca after AV port reversal | 8 hours
change in clearance after AV port reversal | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Willem Boer, MD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost Limburg, Genk, Limburg, Belgium